CLINICAL TRIAL: NCT00596648
Title: A Phase 1b/2 Study of XL184 With or Without Erlotinib in Subjects With Non-Small Cell Lung Cancer
Brief Title: A Study of XL184 (Cabozantinib) With or Without Erlotinib in Subjects With Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XL184-202
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lung Cancer; Non-Small-Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Erlotinib Hydrochloride

ARMS (3):
- Phase 1 Arm (Experimental): Escalating doses of XL184 + erlotinib
  Interventions: Drug: XL184; Drug: erlotinib
- Phase 2 Arm 1 (Experimental): XL184 + erlotinib (dose determined from Phase 1 portion of study)
  Interventions: Drug: XL184; Drug: erlotinib
- Phase 2 Arm 2 (Experimental): XL184 administered as a single agent
  Interventions: Drug: XL184

INTERVENTIONS:
Drug: XL184 — Capsules administered orally daily
Drug: erlotinib — Tablets administered orally daily.
  Arms: Phase 1 Arm; Phase 2 Arm 1

SUMMARY:
The study consisted of a Phase 1 dose escalation/dose de-escalation portion to determine a safe and tolerable combination dose(s) of cabozantinib and erlotinib, and a Phase 2 Simon optimal 2-stage design portion with randomized assignment of subjects in an equal ratio to determine the objective response rate (ORR) of cabozantinib with or without erlotinib in subjects with non-small cell lung cancer (NSCLC) who have progressed after responding to treatment with erlotinib. The doses of cabozantinib used in this study were based on the salt weight, not the freebase weight.

ELIGIBILITY:
Inclusion Criteria-Phase 1:

* Subjects had pathologically confirmed NSCLC and currently have Stage IIIb or IV NSCLC
* Subjects had failed treatment with erlotinib at 150 mg qd
* Subjects had tolerated erlotinib at the dose of the cohort in which they were enrolled (or at a higher dose) for at least 6 weeks (or for the duration of treatment if disease progression had occurred during treatment with erlotinib for less than 6 weeks)
* The subject was at least 18 years old
* The subject had an ECOG performance status of < 2
* The subject had organ and marrow function as follows: - absolute neutrophil count ≥ 1500/mm3, platelets ≥ 100,000/mm3, hemoglobin ≥ 9 g/dL, bilirubin ≤ 1.5 times the upper limit of normal, serum creatinine ≤ 1.5 mg/dL or if serum creatinine > 1.5 mg/dL calculated creatinine clearance ≥ 60 mL/min, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal, amylase and lipase < 1.5 times the upper limit of normal
* Sexually active subjects had to agree to use medically accepted methods of contraception during the course of the study and for 3 months following discontinuation of study treatments (excluding women who are not of child bearing potential and men who have been sterilized)
* Female subjects of childbearing potential had to have a negative pregnancy test at enrollment. Females of childbearing potential were defined as sexually mature women without prior hysterectomy or who had evidence of menses in the past 12 months. However, women who had been amenorrheic for 12 or more months were still considered to be of childbearing potential if the amenorrhea was possibly due to prior chemotherapy, antiestrogens, or ovarian suppression
* The subject had no other diagnosis of malignancy (unless non-melanoma skin cancer, carcinoma in situ of the cervix, or a malignancy diagnosed ≥ 2 years previously, and currently with no evidence of disease)

Exclusion Criteria-Phase 1:

* The subject had received anti-cancer treatment (eg, chemotherapy, radiotherapy, cytokines, or hormones) within 4 weeks with exception of erlotinib (6 weeks for nitrosoureas or mitomycin C) before the first dose of study drug
* The subject had not recovered to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0 Grade ≤1 from clinically significant adverse events (AEs) due to antineoplastic agents, investigational drugs, or other medications that were administered prior to study enrollment
* The subject had symptomatic or uncontrolled brain metastases requiring current treatment, including steroids and anticonvulsants
* The subject had a history of clinically significant hematemesis or a recent history of hemoptysis of > 0.5 teaspoon of red blood or other signs indicative of pulmonary hemorrhage
* The subject had the presence of cavitation, endobronchial lesion or a lesion abutting a major blood vessel
* The subject had serious intercurrent illness, such as uncontrolled hypertension (sustained blood pressure [BP] readings of > 140 mmHg systolic or > 90 mmHg diastolic not controlled with anti-hypertensive medication), unhealed wounds from recent surgery or clinically significant cardiac arrhythmias or a recent history of significant disease such as either symptomatic congestive heart failure or unstable angina pectoris within 3 months or myocardial infarction within 6 months before the first dose of study drug
* The subject was pregnant or breastfeeding
* The subject had an active infection requiring systemic treatment
* The subject had an allergy or hypersensitivity to components of either the cabozantinib or erlotinib formulations
* The subject was incapable of understanding and complying with the protocol or unable to provide informed consent

Inclusion Criteria-Phase 2

* Subjects had pathologically confirmed NSCLC and currently have Stage IIIb or IV NSCLC
* Subjects had: Documented radiological PD, following a prior response, per investigator assessment, to monotherapy with erlotinib, OR; Documented radiological PD, per investigator assessment, following stable disease of at least 6 months on monotherapy with erlotinib
* Subjects who had received subsequent anti-cancer therapy after having progressed on erlotinib (as defined above) also had to have documented radiological PD per investigator assessment to their most recent anti-cancer therapy. If the most recent anti-cancer therapy was erlotinib after having previously progressed on erlotinib (as defined above) the subject also had to have documented radiological PD per investigator assessment to their most recent course of erlotinib
* Subjects had to have tolerated erlotinib at the maximal dose that would be administered in Phase 2 (or at a higher dose) for a minimum of 6 weeks
* Subjects had measurable disease per RECIST
* Subjects had to have 15 unstained consecutive slides of archival or fresh tumor tissue (from one tumor block, frozen tumor tissue, or a paraffin block) identified and designated for shipment to the sponsor if permitted by local regulations (including IRB [Institutional Review Board] policies). The eligibility of subjects with < 15 unstained slides of available archival tissue was discussed with the sponsor
* The subject was at least 18 years old
* The subject had an ECOG performance status of < 1
* The subject had organ and marrow function as follows: absolute neutrophil count ≥ 1500/mm3, platelets ≥ 100,000/mm3, hemoglobin ≥ 9 g/dL, bilirubin ≤ 1.5 times the upper limit of normal, serum creatinine ≤ 1.5 mg/dL or if serum creatinine > 1.5 mg/dL calculated creatinine clearance ≥ 60 mL/min, ALT and AST ≤ 2.5 times the upper limit of normal, amylase and lipase < 1.5 times the upper limit of normal
* Sexually active subjects had to agree to use medically accepted methods of contraception during the course of the study and for 3 months following discontinuation of study treatments (excluding women who are not of child bearing potential and men who have been sterilized)
* Female subjects of childbearing potential had to have a negative pregnancy test at enrollment. Females of childbearing potential were defined as sexually mature women without prior hysterectomy or who had evidence of menses in the past 12 months. However, women who had been amenorrheic for 12 or more months were still considered to be of childbearing potential if the amenorrhea was possibly due to prior chemotherapy, antiestrogens, or ovarian suppression
* The subject had no other diagnosis of malignancy (unless non-melanoma skin cancer, carcinoma in situ of the cervix, or a malignancy diagnosed ≥ 2 years previously, and currently with no evidence of disease)

Exclusion Criteria-Phase 2

* The subject had received: Small molecule inhibitors of vascular endothelial growth factor receptor 2 (VEGFR2)/ kinase insert domain receptor (KDR) at anytime, OR; An investigational anti-cancer agent within 4 weeks of the first dose of study drug, OR; Investigational small molecule inhibitors of EGFR at any time, OR; A small molecule inhibitor of epidermal growth factor (EGF)/EGFR at any time (with the exception of erlotinib and gefitinib), OR; Anti-cancer therapy, including radiation therapy, within 4 weeks of the first dose of study drug (with the exception of gefitinib and erlotinib), OR; Prior therapy with a c-Met inhibitor. Recent (within 3 months) radiation therapy to the thoracic cavity including brachytherapy, unless radiation therapy targeted only bone metastasis
* The subject had not recovered to NCI CTCAE v3.0 Grade ≤1 from clinically significant AEs due to antineoplastic agents, investigational drugs, or other medications that were administered prior to study enrollment
* The subject had symptomatic or uncontrolled brain metastases requiring current treatment, including steroids and anticonvulsants
* The subject had experienced clinically significant hematemesis or hemoptysis of > 0.5 teaspoon of red blood within 3 months before the first dose of study treatment, or other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
* The subject had cavitating pulmonary lesion(s), known endobronchial disease or a pulmonary lesion abutting or encasing a major blood vessel
* The subject had serious intercurrent illness, such as uncontrolled hypertension (sustained BP readings of > 140 mmHg systolic or > 90 mmHg diastolic not controlled with anti hypertensive medication), unhealed wounds from recent surgery or clinically significant cardiac arrhythmias or a recent history of significant disease such as either symptomatic congestive heart failure or unstable angina pectoris within the past 3 months, myocardial infarction, stroke, or transient ischemic attack within the past 6 months
* The subject was pregnant or breastfeeding
* The subject had a clinically significant active infection requiring systemic treatment
* The subject had an allergy or hypersensitivity to components of either the cabozantinib or erlotinib formulations
* The subject was incapable of understanding and complying with the protocol or unable to provide informed consent
* The subject had a history of idiopathic pulmonary fibrosis or interstitial lung disease (ILD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2008-02-12 (Actual); Primary Completion 2012-08-02 (Actual); Study Completion 2012-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Exelixis
Locations (13):
- United States (13):
  - Katmai Oncology Group, Anchorage, Alaska
  - Stanford University Medical Center, Palo Alto, California
  - University of California, Davis, Sacramento, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University/Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - University of Chicago Medical Center, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Park Nicollet Institute, Saint Louis Park, Minnesota
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Case Western Reserve University, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - University of Washington/ Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1-Cohort 1: 75 mg PO qd cabozantinib, 150 mg PO qd erlotinib
- Phase 1-Cohort 2A: 75 mg PO qd cabozantinib, 100 mg PO qd erlotinib
- Phase 1-Cohort 2B: 50 mg PO qd cabozantinib, 150 mg PO qd erlotinib
- Phase 1-Cohort 3A: 125 mg PO qd cabozantinib, 100 mg PO qd erlotinib
- Phase 1-Cohort 4A: 125 mg PO qd cabozantinib, 50 mg PO qd erlotinib
- Phase 2-cabozantinib: single agent cabozantinib 125 mg PO qd
- Phase 2-Cabozantinib + Erlotinib: 125 mg cabozantinib qd and 50 mg erlotinib
Period: Overall Study
Arm/Group | Phase 1-Cohort 1 | Phase 1-Cohort 2A | Phase 1-Cohort 2B | Phase 1-Cohort 3A | Phase 1-Cohort 4A | Phase 2-cabozantinib | Phase 2-Cabozantinib + Erlotinib
Started | 3 | 15 | 17 | 15 | 14 | 15 | 13
Completed | 3 | 14 | 17 | 15 | 14 | 15 | 13
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 2-cabozantinib: cabozantinib single agent 125 mg
- Total: Total of all reporting groups
Arm/Group | Phase 1-Cohort 1 | Phase 1-Cohort 2A | Phase 1-Cohort 2B | Phase 1-Cohort 3A | Phase 1-Cohort 4A | Phase 2-cabozantinib | Phase 2-cabozantinib + Erlotinib | Total
Number analyzed (Participants) | 3 | 15 | 17 | 15 | 14 | 15 | 13 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 8 | 12 | 12 | 7 | 12 | 7 | 60
  >=65 years | 1 | 7 | 5 | 3 | 7 | 3 | 6 | 32
Age, Continuous [Median (Full Range); unit: years] | 56.1 [50 to 79] | 61.6 [30 to 77] | 61.4 [37 to 88] | 57 [35 to 74] | 64.5 [46 to 85] | 54.7 [36 to 74] | 64.8 [44 to 78] | 59.8 [30 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 13 | 10 | 9 | 12 | 7 | 63
  Male | 0 | 6 | 4 | 5 | 5 | 3 | 6 | 29

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Duration of Exposure of Cabozantinib With Erlotinib
Description: Treatment duration was defined as the number of days from the first dose to the last dose (measured in weeks), including any days of treatment interruption that occurred before the last dose of study drug.
Time Frame: From initial dose up to 160 weeks
Population: Safety Population was defined as all participants who received at least one dose of cabozantinib.
Measure: Median (Full Range); unit: Weeks
Groups:
- Phase 1 - Cohort 1: cabozantinib 75mg po QD, plus erlotinib 150mg po QD
- Phase 1 - Cohort 2A: cabozantinib 75mg po QD, plus erlotinib 100mg po QD
- Phase 1 - Cohort 2B: cabozantinib 50mg po QD, plus erlotinib 150mg po QD
- Phase 1 - Cohort 3A: cabozantinib 125mg po QD, plus erlotinib 100mg po QD
- Phase 1 - Cohort 4A: cabozantinib 125mg po QD, plus erlotinib 50mg po QD
Arm/Group | Phase 1 - Cohort 1 | Phase 1 - Cohort 2A | Phase 1 - Cohort 2B | Phase 1 - Cohort 3A | Phase 1 - Cohort 4A
Number analyzed (Participants) | 3 | 15 | 17 | 15 | 14
Weeks
  Cabozantinib (XL184) | 4.43 [3.0 to 7.1] | 8.14 [2.1 to 143.6] | 8.00 [0.4 to 156.7] | 17.00 [6.1 to 80.3] | 20.07 [4.9 to 57.0]
  Erlotinib | 6.57 [5.0 to 9.0] | 10.29 [4.1 to 146.3] | 10.00 [2.4 to 158.7] | 22.00 [8.9 to 84.3] | 22.07 [6.9 to 54.7]

2. Primary Outcome: Phase 2: Objective Response Rate (ORR)
Description: Objective Response Rate is defined as the number of participants for whom the best overall response is complete (CR) or partial response (PR) confirmed by repeat assessments no less than four weeks after the criteria for the initial response were first met.
Time Frame: From initial dose up to 72 weeks
Population: ORR was assessed using the efficacy measurable population.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2 - ARM 1, Cabozantinib ALONE: cabozantinib 125mg po QD
- Phase 2 - ARM 2, Cabozantinib + Erlotinib: cabozantinib po QD 125mg + erlotinib 50mg po QD
Arm/Group | Phase 2 - ARM 1, Cabozantinib ALONE | Phase 2 - ARM 2, Cabozantinib + Erlotinib
Number analyzed (Participants) | 15 | 13
Participants | 1 | 0

3. Secondary Outcome: Phase 2: Duration of Response (DOR) in Participants With a CR or PR
Description: DOR was defined as the time interval from the first documentation of CR or PR to the earlier of the first documentation of definitive disease progression or death from any cause.
Time Frame: From initial dose up to 72 weeks
Population: Safety Population was defined as all participants who received at least one dose of cabozantinib. 'Overall number of participants analyzed' = participants evaluable for this Outcome Measure.
  There were zero responders in Phase 2 - ARM 2, Cabozantinib + Erlotinib arm. So, no data was derived for this endpoint for this arm.
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Phase 2 - ARM 1, Cabozantinib ALONE | Phase 2 - ARM 2, Cabozantinib + Erlotinib
Number analyzed (Participants) | 1 | 0
Weeks | NA [NA to NA] — Per prespecified analysis in the Statistical Analysis Plan, 90% confidence interval was not collected. The DOR for the single participant is not disclosed to protect patient confidentiality. |

4. Secondary Outcome: Phase 2: Progression-Free Survival (PFS)
Description: Progression-free survival is defined as the time from first dose of cabozantinib to disease progression per protocol-defined criteria or death due to any cause, whichever occurs first.
Time Frame: From initial dose up to 72 weeks
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase 2 - ARM 2, Cabozantinib + Erlotinib: cabozantinib 125mg po QD, plus erlotinib 50mg po QD
Arm/Group | Phase 2 - ARM 1, Cabozantinib ALONE | Phase 2 - ARM 2, Cabozantinib + Erlotinib
Number analyzed (Participants) | 15 | 13
months | 1.91 [1.64 to 7.06] | 3.94 [1.54 to 7.26]

ADVERSE EVENTS:
Time Frame: From initial dose through final study visit up to 231 weeks (Phase 1: 159 weeks + Phase 2: 72 weeks)
Description: Safety Population was defined as all participants who received at least one dose of cabozantinib.
Groups:
- Phase 2 - ARM 2, Cabozantinib + Erlotinib: cabozantinib 125mg po QD + erlotinib 50mg po QD
Arm/Group | Phase 1 - Cohort 1 | Phase 1 - Cohort 2A | Phase 1 - Cohort 2B | Phase 1 - Cohort 3A | Phase 1 - Cohort 4A | Phase 2 - ARM 1, Cabozantinib ALONE | Phase 2 - ARM 2, Cabozantinib + Erlotinib
Serious Adverse Events (participants affected / at risk) | 1/3 | 7/15 | 8/17 | 8/15 | 7/14 | 5/15 | 11/13
Other Adverse Events (participants affected / at risk) | 3/3 | 15/15 | 17/17 | 15/15 | 14/14 | 15/15 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 - Cohort 1 (N=3) | Phase 1 - Cohort 2A (N=15) | Phase 1 - Cohort 2B (N=17) | Phase 1 - Cohort 3A (N=15) | Phase 1 - Cohort 4A (N=14) | Phase 2 - ARM 1, Cabozantinib ALONE (N=15) | Phase 2 - ARM 2, Cabozantinib + Erlotinib (N=13)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
GAIT DISTURBANCE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 1 | 2 | 2 | 1 | 1
BRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
BRAIN HERNIATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 3
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
DYSARTHRIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMORRHAGIC STROKE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
INTRAVENTRICULAR HAEMORRHAGE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 2 | 2 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
FATIGUE (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
RECTAL ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OSTENECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 - Cohort 1 (N=3) | Phase 1 - Cohort 2A (N=15) | Phase 1 - Cohort 2B (N=17) | Phase 1 - Cohort 3A (N=15) | Phase 1 - Cohort 4A (N=14) | Phase 2 - ARM 1, Cabozantinib ALONE (N=15) | Phase 2 - ARM 2, Cabozantinib + Erlotinib (N=13)
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 2
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 4 | 1 | 1
ANAEMIA (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2 | 2 | 2 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1 | 2 | 0 | 0
GRANULOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
SPLENIC HAEMORRHAGE (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
TACHYCARDIA (Cardiac disorders) | 0 | 1 | 0 | 2 | 2 | 0 | 0
ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
SUPRAVENTRICULAR BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
SINUS ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
EAR DISCOMFORT (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
HYPOACUSIS (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYPOTHYROIDISM (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
VISION BLURRED (Eye disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 1
DRY EYE (Eye disorders) | 0 | 1 | 2 | 1 | 0 | 1 | 0
EYE DISCHARGE (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
CONJUNCTIVAL OEDEMA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
DIPLOPIA (Eye disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
EYE PRURITUS (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
HALO VISION (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
LACRIMATION INCREASED (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OCULAR ICTERUS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
PHOTOPHOBIA (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 3 | 14 | 13 | 13 | 13 | 9 | 10
NAUSEA (Gastrointestinal disorders) | 2 | 8 | 8 | 12 | 9 | 9 | 7
VOMITING (Gastrointestinal disorders) | 1 | 4 | 8 | 6 | 6 | 5 | 4
CONSTIPATION (Gastrointestinal disorders) | 0 | 2 | 0 | 7 | 5 | 6 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 6 | 2 | 0
DRY MOUTH (Gastrointestinal disorders) | 0 | 1 | 2 | 3 | 4 | 1 | 1
STOMATITIS (Gastrointestinal disorders) | 0 | 1 | 3 | 3 | 3 | 2 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 1 | 4 | 1
DYSPEPSIA (Gastrointestinal disorders) | 1 | 2 | 1 | 3 | 4 | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 3 | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 2 | 0 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 2
FLATULENCE (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 2 | 1 | 0
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0
ORAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 0
ERUCTATION (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1
GLOSSODYNIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
ANORECTAL DISORDER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
CHAPPED LIPS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
GINGIVAL CYST (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
GINGIVAL ERYTHEMA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
GINGIVAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
MOUTH ULCERATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
ORAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
ORAL DISORDER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
ORAL MUCOSAL ERYTHEMA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
PANCREATIC MASS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
PROCTALGIA (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
RETCHING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
SWOLLEN TONGUE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
TONGUE ULCERATION (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
FATIGUE (General disorders) | 3 | 9 | 9 | 10 | 10 | 13 | 10
OEDEMA PERIPHERAL (General disorders) | 0 | 2 | 7 | 1 | 4 | 3 | 3
CHEST PAIN (General disorders) | 0 | 1 | 0 | 0 | 3 | 4 | 1
MUCOSAL INFLAMMATION (General disorders) | 0 | 2 | 0 | 1 | 1 | 1 | 3
ASTHENIA (General disorders) | 1 | 0 | 0 | 1 | 2 | 1 | 0
CHEST DISCOMFORT (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1
CHILLS (General disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0
PAIN (General disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0
PYREXIA (General disorders) | 0 | 1 | 0 | 3 | 0 | 1 | 1
EARLY SATIETY (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
GAIT DISTURBANCE (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
LOCAL SWELLING (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OEDEMA (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
SPINAL PAIN (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
SUPRAPUBIC PAIN (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
XEROSIS (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
SEASONAL ALLERGY (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 3 | 3 | 4 | 1 | 2 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 1 | 1 | 1 | 2 | 1
PARONYCHIA (Infections and infestations) | 0 | 3 | 2 | 2 | 1 | 0 | 1
CANDIDIASIS (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 2 | 0
PHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 1 | 2 | 2 | 2 | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
DIVERTICULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
EYE INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
FUNGAL SKIN INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
HERPES VIRUS INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
LARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
LUNG INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
ORAL HERPES (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
PERIRECTAL ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 0
TRACHEITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 3 | 0 | 1
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
CORNEAL ABRASION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
FACE INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0
TONGUE INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
WOUND (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0
WEIGHT DECREASED (Investigations) | 1 | 6 | 7 | 7 | 7 | 6 | 4
BREATH SOUNDS ABNORMAL (Investigations) | 0 | 2 | 4 | 4 | 2 | 0 | 3
LIPASE INCREASED (Investigations) | 1 | 2 | 3 | 2 | 1 | 4 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 1 | 2 | 1 | 4 | 1
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 | 0 | 2 | 1 | 0 | 2 | 1
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 | 2 | 3 | 3 | 2 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 1 | 1 | 3 | 1 | 1 | 1
BLOOD MAGNESIUM DECREASED (Investigations) | 1 | 2 | 0 | 1 | 2 | 2 | 0
BLOOD PHOSPHORUS DECREASED (Investigations) | 0 | 3 | 1 | 1 | 2 | 1 | 0
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 1 | 1 | 1 | 1 | 1 | 1
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 | 0 | 3 | 0 | 0 | 0 | 0
BLOOD ALBUMIN DECREASED (Investigations) | 0 | 1 | 1 | 0 | 1 | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 1 | 2 | 3 | 0 | 0 | 0 | 0
PLATELET COUNT DECREASED (Investigations) | 1 | 0 | 2 | 0 | 0 | 0 | 1
TRANSAMINASES INCREASED (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 1
AMYLASE INCREASED (Investigations) | 0 | 2 | 0 | 1 | 1 | 1 | 0
BLOOD CHLORIDE DECREASED (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
HAEMOGLOBIN DECREASED (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 1
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 1
PROTHROMBIN TIME PROLONGED (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
BACTERIAL TEST POSITIVE (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
BLOOD BILIRUBIN DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
BLOOD CALCIUM DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
BLOOD CREATINE PHOSPHOKINASE MB INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
BLOOD POTASSIUM DECREASED (Investigations) | 1 | 2 | 1 | 1 | 0 | 0 | 0
BLOOD UREA INCREASED (Investigations) | 1 | 2 | 1 | 0 | 0 | 0 | 0
BLOOD URINE PRESENT (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
CARDIAC MURMUR (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
LYMPH NODE PALPABLE (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
PLATELET COUNT INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
RED CELL DISTRIBUTION WIDTH INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
RESPIRATORY RATE INCREASED (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
SKIN TURGOR DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
URINE LEUKOCYTE ESTERASE POSITIVE (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 7 | 11 | 10 | 11 | 8 | 5
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 5 | 4 | 6 | 3 | 3 | 4
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 2 | 4 | 2 | 6 | 5 | 2 | 4
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 3
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 2 | 2 | 3 | 2 | 1
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 6 | 3 | 1 | 2
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 4 | 1 | 2 | 0 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 1 | 1 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 2 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
HYPERAMYLASAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYPERLIPASAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 3 | 2 | 2 | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 5 | 2 | 1 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 2 | 1 | 2 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3 | 0 | 2 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 2 | 3 | 0 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 3 | 2 | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 2 | 0 | 2 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 3 | 0 | 0 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
DYSGEUSIA (Nervous system disorders) | 0 | 3 | 4 | 8 | 6 | 3 | 3
DIZZINESS (Nervous system disorders) | 0 | 5 | 3 | 6 | 7 | 3 | 1
HEADACHE (Nervous system disorders) | 0 | 3 | 2 | 5 | 4 | 4 | 4
HYPOAESTHESIA (Nervous system disorders) | 0 | 1 | 1 | 1 | 2 | 1 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 1
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 0
DYSKINESIA (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 2 | 1 | 2 | 0 | 0 | 1
SINUS HEADACHE (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
AGEUSIA (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
APHASIA (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
BALANCE DISORDER (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
BRAIN OEDEMA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
BURNING SENSATION (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
COGNITIVE DISORDER (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
CRANIAL NERVE DISORDER (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
DYSARTHRIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
LETHARGY (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
NEURALGIA (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
PRESYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
SPEECH DISORDER (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
TONGUE PARALYSIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
VIITH NERVE PARALYSIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
VISUAL FIELD DEFECT (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 3 | 1 | 2 | 3 | 0
DEPRESSION (Psychiatric disorders) | 0 | 0 | 3 | 1 | 2 | 2 | 0
INSOMNIA (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 4 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 1
ANHEDONIA (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
AGITATION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
DELIRIUM (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HALLUCINATION (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
SLEEP DISORDER (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
SOMNAMBULISM (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
DYSURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
NOCTURIA (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
PROTEINURIA (Renal and urinary disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
AZOTAEMIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
MICTURITION URGENCY (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
BARTHOLIN'S CYST (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
GENITAL LESION (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
GENITAL RASH (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
METRORRHAGIA (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
VULVOVAGINAL PRURITUS (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 6 | 4 | 7 | 4 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 4 | 6 | 8 | 1
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2 | 3 | 1 | 3 | 3
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 2
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 1 | 1 | 0 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 2 | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 2 | 1 | 1 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
RALES (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 1
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OROPHARYNGEAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 9 | 7 | 6 | 4 | 3 | 4
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 2 | 6 | 4
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 | 4 | 1 | 1 | 4 | 6 | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 3 | 2 | 1 | 3
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 3 | 1 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 1 | 1 | 0
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 0
HAIR COLOUR CHANGES (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | 2 | 1 | 0
BLISTER (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
HYPERTRICHOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
NAIL BED TENDERNESS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
SKIN HYPOPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 4 | 0 | 3 | 2 | 3 | 4
HOT FLUSH (Vascular disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0
FLUSHING (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
HYPOTENSION (Vascular disorders) | 0 | 4 | 0 | 3 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes